CLINICAL TRIAL: NCT02069626
Title: The Effect of Compression Time for Secure Stapling With a Linear Stapler in Laparoscopic Gastric Bypass Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, mehmet ali yagci, MD, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013/214
Record Dates: First submitted 2014-02-18; First posted 2014-02-24 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Bleeding of the Staple Line

ARMS (3):
- No wait (Active Comparator): Usage of linear stapler without waiting of compression time
  Interventions: Procedure: compression time of the laparoscopic linear stapler
- 20 second wait (Active Comparator): Usage of linear stapler with 20 second compression time
  Interventions: Procedure: compression time of the laparoscopic linear stapler
- 60 second wait (Active Comparator): Usage of linear stapler with 60 second compression time
  Interventions: Procedure: compression time of the laparoscopic linear stapler

INTERVENTIONS:
Procedure: compression time of the laparoscopic linear stapler

SUMMARY:
Bleeding from the staple line is a complication of linear stapling. After clamping, a short period after firing of the laparoscopic linear stapler is recommended. That is, the clinician should continue to press the tissue between the prongs of the device to achieve adequate hemostasis at the staple line. The significance of the waiting period for hemostasis at the staple line has not been empirically clarified in humans. In this study, the investigators compared the number of bleeding points use of the laparoscopic linear stapler. Consequently, the investigators assessed the effects of time after the firing of linear stapling in patients who underwent laparoscopic gastric bypass.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of morbid obesity
* Must be laparoscopic surgery

Exclusion Criteria:

* Usage of anti-coagulant
* Presence of impaired blood clotting

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Number of the bleeding points at the staple line | intraoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Turgut Özal medical center, Malatya, Malatya, Turkey (Türkiye)